CLINICAL TRIAL: NCT05743400
Title: Thymoglobulin® Pharmacokinetics for Graft-versus Host Disease in Children and Adults Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Thymoglobulin® Pharmacokinetics in Patients Undergoing Hematopoietic Stem Cell Transplantation
Acronym: PHASAL-GA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL21_1186; 2022-501594-39-00 (EU CTIS Number)
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hematopoietic Stem Cell Transplantation-Associated Thrombotic Microangiopathy
Keywords: Hematopoietic stem cell transplantation; Pharmacokinetics; HSCT; Anti-thymocyte globulin; Graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Injections; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental treatment arm (Experimental): Children over two years and adults undergoing a first hematopoietic stem cell transplantation will receiveThymoglobulin® as part of the conditioning.
  Interventions: Drug: Thymoglobulin 25 milligrams (mg) Injection; Biological: blood test

INTERVENTIONS:
Drug: Thymoglobulin 25 milligrams (mg) Injection — Patients will receive thymoglobulin between 5 and 20 milligrams/kilograms (mg/kg) as an intravenous infusion over a period of 2 to 5 days depending on the dose and the transplant package chosen by the physician.
Biological: blood test — Thymoglobulin® serum levels
  Time frame : samples will be drawn at the following points :
  * 1 after each end of perfusion ;
  * 1 though concentration before each perfusion ;
  * 3 blood samples in 3 different days during the first week;
  * 1 weekly for 2 weeks post HSCT.

SUMMARY:
Thymoglobulin is widely applied as serotherapy in order to prevent acute graft-versus-host disease (GvHD) and graft rejection in patients undergoing non-Human Leukocyte Antigen (HLA)-identical hematopoietic stem cell transplantations (HSCT), with a delicate balance between prevention of GvHD and the promotion of immune reconstitution. Thymoglobulin is known as a drug with high pharmacokinetic (PK) variability. This variability influences drug exposure, which in turn determines the drug response of pharmacodynamics (PD). In order to maintain efficacy while reducing adverse effects of drugs across the entire age range, identification of the PK/PD relationships and the effect of growth and maturation on the different PK and PD parameters involved are crucial.

The investigators hypothesise that a better knowledge of Thymoglobulin PK and its covariates would help to individualise dosage regimen and would improve clinical outcomes, such as GvHD and immune reconstitution.

The investigators aim to build a population PK model of Thymoglobulin in order to study PK variability and its covariates. This model will help in optimizing dosage regimen in an individually way.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving Thymoglobulin therapy as part of a first HSCT
* Age ≥ 2 years
* Lansky or karnofsky score ≥ 50%.
* Enrolled in a social security plan
* Patient 18 years of age or older who is informed and has consented to participate in the study or minor patient whose parents/guardians have been informed and have given consent for the minor patient to participate in the study
* Female patients of childbearing potential must have an effective method of contraception (a pregnancy test will also be performed at inclusion).

Exclusion Criteria:

* Patient having received serotherapy (Thymoglobulin® or other) within 3 months before this HSCT
* Patient receiving another serotherapy during conditioning (Campath®)
* Patients with uncontrolled acute or chronic infections for which any form of immunosuppression would be contraindicated
* Known hypersensitivity to Thymoglobulin®.
* Pregnant or lactating women
* Patient participating simultaneously in another study of an investigational drug (no exclusion period)
* Patient under legal protection or deprived of liberty

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) | until elimination tf the drug (maximum 3 weeks post hematopoietic stem cell transplantation)
  Measure of the Thymoglobulin® exposure by the PK criteria : Area under the concentration-time curve (AUC) .
  AUC is measured by day since the first day of Thymoglobulin infusion during conditioning (day 0) until elimination tf the drug. AUC is expressed as milligrams/hour/Liter. (mg/h/L)

SECONDARY OUTCOMES:
Objective function value (OFV) | until elimination tf the drug (maximum 3 weeks post hematopoietic stem cell transplantation)
  Comparison of the OFV of different build population pharmacokinetic models based on results of pharmacokinetic analysis, from start of thymoglobulin® infusion until elimination of the drug
Coefficient of variation of AUC | until elimination tf the drug (maximum 3 weeks post hematopoietic stem cell transplantation)
  Ratio of typical variation of AUC to the mean AUC. AUC is measured by day since the first day of Thymoglobulin infusion during conditioning (day 0) until elimination of the drug

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite